CLINICAL TRIAL: NCT03442348
Title: Utilising Omega 3 and Fibre to Improve Metabolic Health: A Proof of Concept Nutritional Intervention Study Targeting the Gut Microbiome
Brief Title: Omega 3 and Fibre Intervention Study to Improve Metabolic Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 234186
Record Dates: First submitted 2017-10-11; First posted 2018-02-22 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Metabolic Disease; Immune Function; Cardiovascular Diseases; Systemic Inflammation
Keywords: Omega 3; Fibre; Gut microbiome; Metabolic profile; Dietary intervention; Randomised Control Trial
MeSH Terms: conditions — Metabolic Diseases; Cardiovascular Diseases | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Intervention Model Description: The study will be a randomised controlled parallel intervention study in which participants will be grouped into 2 different study arms.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega 3 fatty acid supplements (Experimental): Participants in this arm (N>32) will be required to take one 500mg capsule of Omega 3 along with a meal daily for 6 weeks.
  Interventions: Dietary Supplement: Omega 3 fatty acid
- Inulin fibre (Active Comparator): The participants in the control arm (N>32) will be asked to take 20 g of fibre (inulin fibre) per day for a period of 6 weeks.
  Interventions: Dietary Supplement: Inulin fibre

INTERVENTIONS:
Dietary Supplement: Omega 3 fatty acid — Participants in the bottom median of dietary fibre intake (<15 g per day) will be randomised into one of two arms. Participants in the second arm (N>32) will be required to take one 500mg capsule of Omega 3 along with a meal daily for 6 weeks.
  Arms: Omega 3 fatty acid supplements
Dietary Supplement: Inulin fibre — The participants in the control arm (N>32) will be asked to take 20 g of fibre (resistant starch + inulin) per day that are known favour production of SCFAs in the colon for a period of 6 weeks. The inulin powder will be provided in pre-weighed sachets containing 10g each which can be taken mixed in water or a suitable beverage of choice taken twice (morning and evening) per day.
  Arms: Inulin fibre

SUMMARY:
Metabolic syndrome represents a major health burden worldwide affecting 20-30% of the population. This clustering of abnormalities that confers an increased risk of cardiovascular disease and type 2 diabetes mellitus, is the hallmark of "unhealthy" aging in longevity studies. Preventive strategies have so far failed since they have focused mainly on reducing caloric intake, ignoring the metabolic dysfunction in the aging body. The growing importance of the gut microbiota in all aspects of human health is clear, and unlike our genomes is potentially highly modifiable and tightly related to metabolic and immune efficiency, energy and fatty acid metabolism and satiety hormones. The investigators and others have reported that higher microbiome diversity correlates with significantly lower long-term risk of weight gain and metabolic syndrome. The investigators have recently shown that serum levels of omega-3 fatty acids correlate with higher microbiome diversity, and increased abundance of bacteria that produce butyrate are linked to lower inflammation of the gut. The investigators therefore propose to carry out a proof of concept nutritional intervention study in the TwinsUK cohort. The TwinsUK sample is probably the most detailed omic and phenotypic resource in the world and is ideal for this study. The mechanisms that result in improved microbiome composition and diversity will be explored in a highly focused novel interventional study hypothesizing that key fatty acid pathways are crucially involved in the link between diet, microbiome, immune phenotypes and metabolic syndrome. The specific objectives are to measure changes in gut microbiome composition in response to fibre supplementation compared to omega-3 fatty acid supplementation. The study will measure faecal metabolites relevant to fatty acid metabolism (short chain fatty acids), the abundance of microbial species linked to higher or lower inflammation and immune cell phenotypes to unravel the link between inflammation, diet and metabolic syndrome. There is a real lack of good diet intervention studies in this field and if successful this trial will pave the way to funding a wide variety of other diet intervention studies.

DETAILED DESCRIPTION:
Diet and nutrition are key determinants of chronic disease. However, additional information is needed on which bioactive compounds and in what amounts they should be consumed to obtain a given health benefit. One of the biggest recent breakthroughs in science has been realisation of the importance of the contents, function and homeostasis of the gut microbiome in human health.

Dietary fibre: The influence of diet on the microbiome is illustrated by vast differences across cultures where African communities who have a plant based diet consume 7-fold more fibre compared with the West obtaining more of their energy requirements via utilization of gut microbiota. Hunter-gatherers have been shown to have 30-40% greater numbers and diversity of species than Western populations. Also, a multigenerational murine study showed a Western diet was responsible for depletion of microbiota diversity. Diversity is emerging as the common marker of good gut health across populations and related to production of beneficial short chain fatty acids (SCFAs). The fermentation of dietary fibre changes the profile of microbial-derived metabolites within the GI tract, most importantly SCFAs. Low fibre intake results in reduced production of SCFAs and also shifts the gastrointestinal (GI) microbiota metabolism to the utilization of less favourable nutrients, leading to the production of potentially detrimental metabolites derived from the fermentation of amino acids. Prevention of the generation of such metabolites through dietary fibre is one of the main mechanisms for the prevention of colon cancer. There is considerable observational evidence that fibre intake is beneficial for human health from observational epidemiological studies. However, findings from intervention studies are less consistent. The variability in human intervention studies could also arise from the highly inter-individualized responses of the human GI microbiome to dietary fibres providing a rationale for the individualization of dietary fibre applications.

Omega 3 fatty acids: In humans, omega-3 fatty acids are readily incorporated into cell membranes resulting in increased cell fluidity, which may improve glucose transport. Additionally, omega-3 supplementation enhances resting fat oxidation and glycogen storage, potentially contributing to improved insulin sensitivity. Omega-3 supplementation may also reduce cardiovascular disease risk by reducing circulating very-low-density lipoproteins (LDL), triacylglycerols and free fatty acids (FFA). It also has additional anti-inflammatory and antithrombotic properties. Previously published data by the investigators suggest the potential use of omega-3 supplementation to improve the microbiome composition. Although trials of supplements are inconsistent, current recommended daily intake for omega-3 is 250 mg (active EPA and DHA) for the general population and higher for patients with cardiovascular disease.

The study will be a proof of concept mechanistic study that will show to what extent omega-3 fatty acid supplementation adds to the benefits of a probiotic intervention in terms both of microbiome diversity and composition and of SCFA production. Moreover, it will show whether this results in measurable improvements in other markers of fatty acid metabolism and in the balance of various T-cell lineages some of which are pro-inflammatory and others which are anti-inflammatory. In this study we will test if 1) intake of fibre induces an increase in microbiome diversity, increased SCFA production in the gut and less inflammatory T-cell composition 2) omega-3 supplementation provides a comparable benefit in terms of microbiome diversity and cardiometabolic improvement to that supplied by fibre.

The study will be a randomised controlled intervention study in which participants will be grouped into two different treatment arms. Randomisation will control for equal distribution of key characteristics that may confound between group comparisons and will be assessed by analysis of baseline data.

80 participants over the age of 18 years will be recruited from the TwinsUK database.The total length of the dietary intervention will be 6 weeks with an initial visit at baseline, and one final visit at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant eligibility includes those aged >18 years who have a body mass index (BMI) between 20 and 39.9 kg/m2. Participants must have low habitual fibre consumption of less than 15g/day.

Exclusion Criteria:

* Refuse or are unable to give informed consent to participate in the study
* Consume on average >15 g/day of NSP and RS (men and women) as part of their diets
* Are taking the following medications: immunosuppressants, amiodarone and/or perhexiline
* Are currently following or anticipated to commence a specialised commercially available weight loss diet and/or program
* Have a diagnosis of insulin dependent diabetes mellitus
* Have a current or prior history of cardiovascular, cerebrovascular or peripheral vascular disease
* Have clinically relevant pulmonary, gastro-intestinal, renal, metabolic, hematological, neurological, psychiatric, systemic or any acute infectious disease or signs of acute illness
* Are women who are pregnant
* Have psychosocial or gastrointestinal (e.g. malabsorptive conditions such as IBS, coeliac)
* Have contraindications included bulimia nervosa, substance abuse, clinically significant depression, or current psychiatric care
* Have had a recent (within 3 months) of change in dose/regime or introduction of vitamin E, C or high dose vitamin D (>3000 IU), fish oil, prebiotics or probiotics.
* Are vegetarian and thus unwilling to take fish oil capsules
* People on anticoagulants and people with atrial fibrillation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome diversity | 3-6 weeks
  16s sequencing will be carried out on whole stool samples to measure gut microbial diversity and composition. Stool samples collected and frozen within two hours will be assessed in greater detail for markers of microbiome function and gut health which include measuring key short-chain fatty acids using mass spectrometry.
Metabolites | 3-6 months
  Measure of faecal metabolites such as short chain fatty acids, blood glucose, blood lipids, ketone bodies
Immune phenotypes | 3-6 months
  Markers of immune response measured using peripheral blood mononuclear cells

SECONDARY OUTCOMES:
Assessment of hunger | 6 weeks
  Appetite questionnaire
Assessment of sleep | 6 weeks
  Sleep pattern will be assessed using a validated questionnaire (Medical Outcomes Survey sleep questionnaire) at baseline, mid-intervention and the end of the intervention.
Assessment of physical exercise | 6 weeks
  Physical exercise will be assessed using a validated questionnaire(Sf-12) at baseline, mid-intervention and the end of the intervention.
Assessment of Mood | 6 weeks
  Mood will be assessed using a validated questionnaire (HADS, anxiety and depression validated questionnaire) at baseline, mid-intervention and the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Valdez, Dr, Principal Investigator — King's College London
Locations (1):
- King's College London, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided